CLINICAL TRIAL: NCT02188017
Title: ACTHAR Gel for Chronic Pulmonary Sarcoidosis (ACPS)
Acronym: ACPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Robert P Baughman, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACPS
Record Dates: First submitted 2014-04-24; First posted 2014-07-11 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis; Pulmonary Sarcoidosis
Keywords: prednisone, methotrexate, sarcoidosis, azathioprine
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 80 units (Active Comparator): 80 units ACTHAR gel will be given twice a week for 22 weeks after initial loading
  Interventions: Drug: Acthar gel
- 40 units (Active Comparator): 40 units of ACTHAR gel will be given twice a week for 22 weeks after loading
  Interventions: Drug: Acthar gel

INTERVENTIONS:
Drug: Acthar gel — Given 80 units daily for 10 days, then randomized to receive either 40 or 80 units twice a week
  Other Names: ACTH; Cortysin

SUMMARY:
An randomized trial of two maintenance doses of Acthar Gel for patients with chronic pulmonary sarcoidosis. Patients will be observed for 24 weeks of treatment.

DETAILED DESCRIPTION:
This is a multi-center double-blind trial to determine dose and effect size. A total of 20 chronic pulmonary sarcoidosis patients will be recruited at eight clinical sites across the United States.

After initial evaluation, including pulmonary function, CT and PET scanning, patients will be randomized to receive 80 Units if Acthar gel daily for 10days, followed by either 40 or 80 units of Acthar gel twice a week for an additional 22 weeks.

At the end of total 24 weeks of treatment, they will undergo repeat evaluation including pulmonary function, CT, and PET scanning.

ELIGIBILITY:
Inclusion Criteria:

* Patient with biopsy confirmed sarcoidosis meeting American Thoracic Society criteria 23
* Patient on >5 mg prednisone for pulmonary indications
* FVC <85% predicted
* Prednisone dose not reduced in prior 3 months
* Deterioration of pulmonary disease over the past year
* Decrease in FVC >5%
* Age: 18 through 90 (i.e., candidates must have had their 18th birthday, but not had their 91st birthday).

Exclusion Criteria:

adrenal insufficiency (Addison's disease)

* Scleroderma
* a fungal infection
* herpes infection of the eyes
* osteoporosis
* a stomach ulcer
* congestive heart failure
* high blood pressure
* recent surgery
* if you are allergic to pork proteins
* Do not receive a smallpox vaccine or any "live" vaccine while you are using corticotropin.
* Patients receiving anti-Tumor Necrosis Factor antibody (e.g. infliximab, adalimumab) in prior six months
* Uncontrolled diabetes, hypertension, or other contra-indication to increased dosage of glucocorticoids
* Patients requiring therapy for pulmonary hypertension
* Females of childbearing potential who are known to be pregnant and/or lactating or who have a positive urine pregnancy test on screening.
* Current participation in another research drug treatment protocol (patient cannot start another experimental agent until after 90 days)
* Any other condition that the investigator feels would pose a significant hazard to the patient if Acthar Gel therapy is initiated.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Steroid toxicity | 24 weeks
  Cumulative toxicity between two arms of study over 24 weeks of study This will be assessed using a steroid toxicity questionnaire

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 24 weeks
  Change in FVC over course of study
Chest x-ray | 24 weeks
  Change in chest x-ray
PET scan | 24 weeks
  Change in lung uptake of PET scan during course of study
Sarcoidosis Health Questionnaire | 24 weeks
  Change in quality of life as assessed by King's Sarcoidosis Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Baughman RP, Sweiss N, Keijsers R, Birring SS, Shipley R, Saketkoo LA, Lower EE. Repository corticotropin for Chronic Pulmonary Sarcoidosis. Lung. 2017 Jun;195(3):313-322. doi: 10.1007/s00408-017-9994-4. Epub 2017 Mar 28. PMID 28353116